CLINICAL TRIAL: NCT04017143
Title: Multi-Level Communication Strategies for HPV Vaccination in Hmong Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00002064
Record Dates: First submitted 2018-12-17; First posted 2019-07-12 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: HPV-associated Cancer

STUDY DESIGN:
Intervention Model Description: Two-Arm Randomized Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV App group (Experimental): Participants will be assigned to receive an HPV app.
  Interventions: Behavioral: HPV app intervention
- Usual Care (No Intervention): This is a usual care group that receives a brochure that is usually distributed by a clinic.

INTERVENTIONS:
Behavioral: HPV app intervention — Participants assigned to this group will receive an HPV app that targets a dyad of parent and a teen boy or girl.
  Arms: HPV App group

SUMMARY:
The specific aims are: 1) to design a multilevel, theory-driven, highly interactive, culturally and cognitively tailored hAppy app intervention to facilitate HPV vaccination completion among Hmong adolescents and their parents using CBPAR; 2) establish a systematic health care provider protocol for identifying and engaging Hmong adolescents and their parents in the use of the hAppy app; and 3) examine participants' intent, knowledge and self-efficacy of HPV vaccinations, perceptions of the hAppy app and their patient-provider experiences. This study will advance existing knowledge of mHealth's impact on populations at risk for cancer and contribute new, important information to cancer health disparities research. If found to be effective, this intervention will have extensive implications for prevention of other types of cancer among different underserved populations, potentially reducing cancer-related disparities, morbidity, and mortality.

DETAILED DESCRIPTION:
A quarter million Hmong Americans (Hmong) reside in the United States and 25% live in the Twin Cities metropolitan area. With a median age of 20.4 years old, this young community has a poverty rate of 26% in Minnesota and 27.4% nationally. Cervical cancer knowledge and prevention, such as awareness of HPV's effectiveness in reducing cancer risk, is low among Hmong women (19-50%) and men (38%), which may explain Hmong's high cervical cancer incidence rates (three times higher than other Asian Americans (AA) and four times higher than Non-Hispanic Whites). This problem is further aggravated by the rise of cervical cancer incidence and mortality rates among Hmong women. Clearly, multilevel strategies to increase HPV vaccination rates and reduce HPV-related cancers among Hmong are urgently needed. Yet Hmong women face structural and cultural barriers that limit their access to preventive health care. Language difficulties, poor health literacy, lack of time or transportation, visiting a doctor only when symptomatic or in pain and abstaining from gynecological visits due to embarrassment are some of these barriers. These barriers and beliefs must be carefully integrated into the design of any effective multilevel strategy to promote HPV vaccination uptake and completion. This study proposes to use a Community-Based Participatory Action Research (CBPAR) approach to develop and test the effectiveness of a theory-based culturally and cognitively appropriate mobile application (hAppy app) intervention that facilitate HPV vaccination completion among Hmong adolescents (11 to 17 years old) and their parents. Mobile health (mHealth) technology is a promising tool allowing for effective person-centered customization. The study's primary objective is to evaluate the effectiveness of hAppy app intervention in Hmong adolescents and their parents. 100 Hmong adolescents and their parents will be recruited and a single blind, two arm, randomized controlled trial will be conducted. Participants will be randomized by a 1:1 ratio to receive the hAppy app intervention (N=50) or usual care (UC, N=50) for a 9-month period.

ELIGIBILITY:
Inclusion Criteria:

* Teen: (1) aged between 11-17, (2) not yet completed HPV vaccination, (3) living in Minnesota
* Parents: those who have teen child aged between 11-17

Exclusion Criteria:

* Teens who have completed HPV vaccination

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of HPV vaccination (completion of recommended HPV vaccine) | 9-months
  Number of teen participants who receive the complete series of recommended HPV vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Twin Cities, Minneapolis, Minnesota, United States